CLINICAL TRIAL: NCT03120039
Title: Measuring Upper Extremity Functional Movement with Accelerometry: FitBit Vs Actigraph
Brief Title: Measuring Upper Extremity Functional Movement with Accelerometry: FitBit® Vs Actigraph®
Status: Completed | Type: Observational
Sponsor: Rowe, Veronica, M.D. (Individual)
Responsible Party: Principal Investigator, Veronica Rowe, Assistant Professor, Rowe, Veronica, M.D.
Other Study IDs: FitBit vs Actigraph
Record Dates: First submitted 2017-04-11; First posted 2017-04-19 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2017-04

CONDITIONS: Motor Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy adults: Healthy adults without any limitations in upper extremity movement or function.

SUMMARY:
To determine the criterion validity of the FitBit® Flex™ compared to the ActiGraph's Bluetooth® Smart wGT3X-BT wireless activity monitor, and contribute to the clinical utility of accelerometry measurement of UE movement.

DETAILED DESCRIPTION:
Participants will wear two different accelerometers (FitBit and Actigraph) to record normal, everyday movement. Data from each accelerometer will be compared to determine similarity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults with no upper extremity limitations

Exclusion Criteria:

* Upper extremity limitations

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-05-01 (Actual)

PRIMARY OUTCOMES:
Steps | 24 hours
  Number of steps

IPD SHARING:
Plan to Share IPD: No